CLINICAL TRIAL: NCT05850390
Title: Real-time Remote Asthma Monitoring Through Smartphone Voice Analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sonde Health (Industry)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SH2021.ASTHMA01
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosed asthma patients: Adults aged 18 and above who have been diagnosed with persistent asthma or allergy with asthma as a co-morbidity and are prescribed a controller medication.
  Interventions: Other: Respiratory-Responsive Vocal Biomarker application

INTERVENTIONS:
Other: Respiratory-Responsive Vocal Biomarker application — A smartphone app that allows participants to receive a respiratory-responsive vocal biomarker (RRVB) score by recording a 6-second held "ahh" vowel elicitation. The applications returns the RRVB score which has previously been validated to correspond to the likelihood that the user's voice is similar to those of people diagnosed with asthma. This study will examine if the RRVB scores correlate with respiratory function and symptoms in asthma patients.

SUMMARY:
This study examines the impact of home-based monitoring of respiratory function in asthma patients via a smartphone-based vocal biomarker platform. Previous work from cross-sectional studies has indicated that brief voice samples, analyzed by machine learning models, can predict the presence of respiratory conditions (asthma, COPD, ILD, COVID-19 and persistent cough) with an accuracy of approximately 70%. The present study seeks to extend these findings to establish whether the same vocal biomarker models can accurately track changes in respiratory function in asthma patients, and whether this capability, when incorporated into a smartphone app similar to those used for home-based asthma management, can improve relative level of asthma control.

DETAILED DESCRIPTION:
The study aims to investigate whether home-based monitoring of respiratory function in asthma patients using a smartphone-based vocal biomarker platform can improve the level of asthma control. The study will involve 70 patients aged 18 years and above with a primary diagnosis of asthma or allergy with asthma as a comorbidity, with an Asthma Control Test (ACT) score of less than or equal to 19 at baseline. The primary objective of the study is to assess whether vocal biomarker scores can provide asthma patients with real-time objective information on their respiratory function using voice samples recorded on their personal smartphone device.

The secondary objectives of the study include determining whether smartphone apps incorporating vocal biomarker capabilities can improve asthma control, assessing patient engagement with the apps, and examining the impact of the apps on healthcare utilization in asthma patients. Exploratory objectives include determining how the participant's digital health literacy phenotype can assist in creating engagement with asthma management apps and developing care team dashboards for providers to assist in periodic evaluation of patient status using a vocal biomarker platform.

The study will explore voice recordings for potential new machine learning model development to assess whether different vocal biomarker combinations can provide superior respiratory function monitoring ability than the established Respiratory Symptom Risk scores that were developed from cross-sectional asthma data. The primary endpoints of the study are performance-related measures of Respiratory Symptom Risk score, and the secondary endpoints include the proportion of subjects with ACT improvement and the proportion of participants providing voice samples.

The study will be conducted for three months in clinics providing care to asthma patients, typically asthma/allergy clinics. The Sonde Health App will be used to provide vocal biomarker respiratory symptom risk scores to patients on their personal smartphone device and be used for data collection. The findings of the study could help establish whether the same vocal biomarker models can accurately track changes in respiratory function in asthma patients and whether incorporating this capability into smartphone apps can improve the level of asthma control.

ELIGIBILITY:
Inclusion Criteria:

1. Own an eligible smartphone (iOS or Android) that is able to download and run the Sonde Health app
2. Willing to sign up for a Sonde app account
3. Agreement with the subject consent information presented on the Sonde app.
4. Stated willingness and ability to comply with all study procedures for the duration of the study
5. Male or female, aged 18 or above
6. Able to read and speak English (required to follow app instructions and provide correct voice elicitations)
7. Pregnant women are allowed to participate
8. Have a medical diagnosis of persistent asthma, or allergy with asthma as a co-morbidity, and a prescribed controller medication
9. ACT score <= 19 on day of enrollment
10. New or existing patients are eligible
11. Asthma and COPD as comorbidities are allowed

Exclusion Criteria:

1. Speech disorder or impediment (clinician judgment)
2. Difficulties reading or responding to instructions and questions on a smartphone screen
3. End-stage COPD or other condition requiring home oxygen
4. Anticipated inability to conduct daily peak flow meter readings at home
5. Participation in asthma-focused medication studies or trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is testing the use of the Sonde Health app in patients with persistent asthma or allergy with asthma as a co-morbidity who are prescribed controller medication. Participants must be 18 or older, speak English, and have an eligible smartphone. Daily peak flow meter readings are required. New or existing patients and pregnant women can participate. No speech disorders, smartphone issues, or end-stage COPD. No ongoing asthma trials.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
RRVB monitoring performance vs. PEF | Enrollment through end of month 3
  Sensitivity, specificity and odds ratio of RRVB score to identify peak flow scores vs. personal best in green (>=80%, G), yellow (>=50%, <80%, Y) and red zones (<50%, R)

SECONDARY OUTCOMES:
ACT improvement | End of month 1, 2 and 3
  The proportion of participants with ACT improvement >=3 points
RRVB tool engagement | During month 1, 2, and 3
  The proportion of participants providing voice samples on =>50% days

CONTACTS AND LOCATIONS:
Overall Officials: Sunit P Jariwala, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen E, Song X, Joachim D, Ch'en PY, M Green S, Hunt E, Kaur S, Nag R, Pisani O, Thomas S, Adewunmi V, Lutz C, Baghizadeh-Toosi B, Feldman JM, Jariwala S. Respiratory-Responsive Vocal Biomarker for Asthma Exacerbation Monitoring: Prospective Cohort Study. J Med Internet Res. 2025 Sep 23;27:e68741. doi: 10.2196/68741. PMID 40986855